CLINICAL TRIAL: NCT00323414
Title: Randomized Controlled Trial of Omega-3 Fatty Acids in the Treatment of Non-Alcoholic Steatohepatitis in Patients With Type 2 Diabetes Mellitus
Brief Title: Polyunsaturated Fatty Acids (PUFA) in Diabetic Fatty Liver
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DK61732; U01DK061732 (NIH)
Record Dates: First submitted 2006-05-05; First posted 2006-05-09 (Estimated); Results first posted 2018-02-23 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2017-10

CONDITIONS: Fatty Liver
Keywords: PUFA; NASH; Fatty Liver; Insulin resistance; Metabolic syndrome; Nonalcoholic fatty liver disease; Nonalcoholic steatohepatitis; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Fatty Liver; Insulin Resistance; Metabolic Syndrome; Non-alcoholic Fatty Liver Disease; Diabetes Mellitus, Type 2 | interventions — Fatty Acids, Unsaturated; Fish Oils; Corn Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Polyunsaturated fatty acid (Opti-EPA) (Active Comparator): Polyunsaturated fatty acid will consist of purified EPA:DHA (360 mg EPA and 240 mg DHA) 6 gelcaps-3 capsules by mouth 2x per day x 48 weeks
  Interventions: Drug: Polyunsaturated fatty acid (Opti-EPA)
- Placebo (Placebo Comparator): Gelcaps containing corn oil as placebo 6 capsules 3 capsules by mouth 2 x per day for 48 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Polyunsaturated fatty acid (Opti-EPA) — Active experimental arm to patients with diabetes mellitus and non alcoholic steatohepatitis: Eicosapentaenoic acid (EPA):Docosahexaenoic acid (DHA)[360 mg EPA and 240 DHA in each capsule] 6 capsules-3 capsules by mouth 2 x per day x 48 weeks
  Other Names: Fish oil
  Arms: Polyunsaturated fatty acid (Opti-EPA)
Drug: Placebo — Placebo gelcaps containing corn oil identical to the PUFA gelcaps 6 capsules-3 capsules by mouth 2x per day x 48 weeks
  Other Names: Corn oil
  Arms: Placebo

SUMMARY:
Non-alcoholic steatohepatitis (NASH), the most severe form of liver injury in the spectrum of non-alcoholic fatty liver disease (NAFLD), has emerged as the major cause of chronic liver disease in developed countries. Among adults in the United States, the prevalence is between 5.7% and 17%. These rates are expected to increase concurrent with the epidemics of obesity and type 2 diabetes mellitus, which are the major risk factors for NAFLD and NASH. In addition to its high prevalence, NASH is also a progressive fibrotic disease that advances to cirrhosis and liver related death in 20% and 12% of patients, respectively. Among NASH patients with cirrhosis, 40% have liver related death. Diabetics are particularly prone to experience these poor outcomes. No therapy has been proven effective for patients with NASH.

The purpose of this study is to find out whether treatment with polyunsaturated fatty acids (eicosapentaenoic acid [EPA] combined with docosahexaenoic acid [DHA] called Opti-EPA) improves NASH compared to treatment with placebo pills. The placebo pills will contain corn oil and will be contained in a capsule, but have no medical effect on the body. The investigators will determine improvement in NASH from microscopic changes in the subject's liver tissue during 48 weeks of treatment. This means that the subject will need to have a liver biopsy before and after the treatment.

Omega-3 fatty acids are a form of polyunsaturated fats, one of the four basic types of fat that the body gets from food. (Cholesterol, saturated fat, and monounsaturated fat are the others.) One's body does not make this type of fat; it comes from food sources. These fats are found in foods like cold water fish (tuna, salmon, and mackerel), and vegetable products like flaxseed oil and walnuts.

Research shows that polyunsaturated fats are good for people. Studies have shown that it is good for heart health by playing a role in keeping blood cholesterol levels low, keeping irregular heart rhythms stable, and reducing blood pressure.

The drug being studied, Opti-EPA, is a nutritional supplement. They do not have to be reviewed by the Food and Drug Administration (FDA) like medicines do. Opti-EPA is considered experimental in this study. This means that the United States Food and Drug Administration (FDA) has not approved it for use in people with nonalcoholic fatty liver disease.

DETAILED DESCRIPTION:
Although there is no proven effective treatment of NASH, dietary supplementation with long chain omega-3 polyunsaturated fatty acids (PUFA's) may be beneficial. This suggestion is based on three previously reported observations: first, patients with NASH consume less PUFAs and more saturated fats than subjects without NASH. Second, PUFAs are beneficial in patients with hypertension and hypertriglyceridemia. Third, PUFAs decrease lipid peroxidation and ameliorate hepatic steatosis in animal models of NAFLD.

We therefore hypothesize that the administration of these PUFAs, eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA) will reduce hepatic fat content, inflammation and hepatic injury in patients with type 2 diabetes mellitus who have NASH.

Aims

To determine in patients with type 2 diabetes mellitus who have NASH if dietary supplementation with purified omega-3 fatty acids (EPA and DHA) will:

1. Decrease the histologic severity of NASH.
2. Alter the expression of genes important in the pathways of hepatic lipid synthesis and oxidation.

Study design:

Patients who meet the inclusion criteria will be randomized to receive omega-3 fatty acids or placebo. Stratified randomization will be done based on the NASH Clinical Research Network pathology score of 5.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age >18 years)
* Have type 2 diabetes mellitus with good control of blood sugar (hemoglobin A1c [HbA1c] <7.5%) and will have been on a stable regimen of anti-diabetic agents for more than 4 months.
* NASH established on liver biopsy done within 6 months prior to inclusion in the study as determined by established histologic criteria

Exclusion Criteria:

* Cirrhosis of the liver
* End stage target organ damage in diabetes mellitus: advanced renal failure (serum creatinine > 2.0 mg/dl) with or without dialysis, severe neuropathy, or advanced peripheral vascular disease.
* Any organ dysfunction with anticipated life expectancy of less than 2 years
* Co-existent etiologies for liver disease
* Significant alcohol consumption, defined as more than 30 g per day in men and more than 20 g per day in women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2006-04; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arthur J. McCullough, M.D., Principal Investigator — MetroHealth Medical Center; Srinivasan Dasarathy, M.D., Principal Investigator — The Cleveland Clinic
Locations (2):
- United States (2):
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio

REFERENCES:
- [Background] Younossi ZM, Gramlich T, Matteoni CA, Boparai N, McCullough AJ. Nonalcoholic fatty liver disease in patients with type 2 diabetes. Clin Gastroenterol Hepatol. 2004 Mar;2(3):262-5. doi: 10.1016/s1542-3565(04)00014-x. PMID 15017611
- [Derived] Dasarathy S, Dasarathy J, Khiyami A, Yerian L, Hawkins C, Sargent R, McCullough AJ. Double-blind randomized placebo-controlled clinical trial of omega 3 fatty acids for the treatment of diabetic patients with nonalcoholic steatohepatitis. J Clin Gastroenterol. 2015 Feb;49(2):137-44. doi: 10.1097/MCG.0000000000000099. PMID 24583757

RESULTS

PARTICIPANT FLOW:
Groups:
- PUFA: Purified EPA:DHA (360 mg EPA and 240 mg DHA) 6 gelcaps 3 capsules by mouth 2x per day x 48 weeks
Period: Overall Study
Arm/Group | PUFA | Placebo
Started | 18 | 19
Completed | 18 | 18
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PUFA | Placebo | Total
Number analyzed (Participants) | 18 | 19 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 19 | 37
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 17 | 29
  Male | 6 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Improvement of >= 2 Points in NAFLD Activity Score (NAS)
Description: The non-alcoholic fatty liver disease (NAFLD) activity score (NAS) is a score based on the liver biopsy. It represents the sum of scores for steatosis, lobular inflammation, and ballooning, and ranges from 0-8, with high scores indicating more activity.
Time Frame: 48 weeks
Measure: Count of Participants; unit: Participants
Groups:
- PUFA: Active treatment with PUFA
- Placebo: Placebo arm of therapy
Arm/Group | PUFA | Placebo
Number analyzed (Participants) | 18 | 19
Participants | 8 | 9

2. Secondary Outcome: Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) Values
Description: Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) measures insulin resistance, calculated by fasting insulin (μU/mL) multiplied by fasting glucose (mg/dL), and divided by a constant (405). A higher score indicates higher insulin resistance.
Time Frame: 48 weeks
Measure: Mean (Standard Deviation); unit: HOMA-IR index
Arm/Group | PUFA | Placebo
Number analyzed (Participants) | 18 | 19
HOMA-IR index | 16.1 (10.3) | 13.1 (7.3)

3. Secondary Outcome: Aspartate Amino Transferase (AST) Levels
Description: Aspartate amino transferase (IU/dL) at 48 weeks
Time Frame: 48 weeks
Measure: Mean (Standard Deviation); unit: IU/dL
Arm/Group | PUFA | Placebo
Number analyzed (Participants) | 18 | 19
IU/dL | 41.7 (17.4) | 47.9 (38.1)

4. Secondary Outcome: Alanine Amino Transferase (ALT) Levels
Description: Alanine amino transferase (IU/dL) ay 48 weeks
Time Frame: 48 weeks
Measure: Mean (Standard Deviation); unit: IU/dL
Arm/Group | PUFA | Placebo
Number analyzed (Participants) | 18 | 19
IU/dL | 56.9 (30.9) | 59.6 (43.8)

5. Secondary Outcome: Blood Glucose Levels
Description: Fasting blood glucose
Time Frame: 48 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | PUFA | Placebo
Number analyzed (Participants) | 18 | 19
mg/dL | 150.4 (43.7) | 123.5 (22.9)

6. Secondary Outcome: HbA1C Levels
Description: Hemoglobin A1c
Time Frame: 48 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | PUFA | Placebo
Number analyzed (Participants) | 18 | 19
mg/dL | 7.5 (2.2) | 6.9 (1.1)

ADVERSE EVENTS:
Time Frame: 48 weeks
Description: Patient reported adverse events and abnormal laboratory tests were collected
Arm/Group | PUFA | Placebo
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/18 | 2/19
Other Adverse Events (participants affected / at risk) | 1/18 | 0/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PUFA (N=18) | Placebo (N=19)
Post liver biopsy pain (Surgical and medical procedures) | 0 (0) | 1 (1) — End of treatment, post liver biopsy bleeding requiring blood transfusion in one and none in the other. Both patients showed evidence of perihepatic hematoma and were discharged home uneventfully
Post liver biopsy bleeding (Surgical and medical procedures) | 0 (0) | 1 (1) — Needed 2 units blood transfusion. Discharged uneventfully and is being followed in the clinic subsequently
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PUFA (N=18) | Placebo (N=19)
No tissue (Surgical and medical procedures) | 1 (1) | 0 (0) — Liver biopsy did not yield tissue

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes